CLINICAL TRIAL: NCT04611165
Title: A Phase II Study of Concurrent Nivolumab and External Beam Radiation Therapy for Patients With Advanced Hepatocellular Carcinoma Who Have Vascular Invasion With or Without Sorafenib-Experience in an HBV-endemic Area
Brief Title: Concurrent Nivolumab and External Beam Radiation Therapy for Patients With Advanced HCC
Acronym: Nextrah
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joong-Won Park, Principal Investigator, Clinical Professor, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2019-0274
Record Dates: First submitted 2020-09-28; First posted 2020-11-02 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: External Beam Radiation Therapy; Advanced Hepatocellular Carcinoma Who Have Vascular Invasion; Nivolumab
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single (Experimental): Nivolumab 3mg/kg IV is administered as 30-minute IV infusion every 2 weeks.
  Prescription dose to PTVs as according to the following schema:
  PTV1: 30 - 50 Gy /10 fx, 5Gy fraction dose, 5 days/week (The prescribed dose to PTV will be decided by physician depending on the dose-volume histogram (DVH) constraints of the normal tissues, such as liver, bowel, etc. The detail of DVH constraints of normal tissues are summarized in the following table) PTV2: 30 Gy /10 fx, 3Gy fraction dose, 5 days/week
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — * Nivolumab 3mg/kg IV is administered as 30-minute IV infusion every 2 weeks.
  * EBRT begins 2-7 days after the first dose of nivolumab.
  * The follow-up phase begins when the decision to discontinue study is made. The follow-up phase is defined as the day after the end of study treatment until the day the subject dies.
  Other Names: EBRT

SUMMARY:
To investigate the efficacy and safety of nivolumab for patients with advanced HCC undergoing EBRT

DETAILED DESCRIPTION:
<Treatment phase> Nivolumab 3mg/kg IV is administered as 30-minute IV infusion every 2 weeks. External beam radiotherapy begins 2-7 days after the first dose of nivolumab. The study drug is continued until disease progression, unacceptable toxicity, withdrawal of consent or study closure.

<Follow-Up phase > After the treatment phase, subjects will undergo follow up for survival every 12 weeks (± 7 days) from the last dose or the use of other anticancer treatments and/or therapies, and the survival follow up will be performed for at least 18 months after the enrollment of the last subject. The patient will be followed for survival follow up and the use of other anticancer treatments and/or therapies.

Based on the assumed dropout rate of 12%, a total of 50 subjects need to perform the study (50=44/(1-0.12))

ELIGIBILITY:
Inclusion Criteria:

* Patients with HCC meeting all of following criteria;

  1. Signed written informed consent
  2. Age >= 20
  3. Histological or clinical diagnosis of HCC based on the guidelines of the Korean Liver Cancer Association-National Cancer Center17
  4. Having at least one typical enhanced measurable index lesion (in the liver) by dynamic CT or dynamic contrast-enhanced MRI
  5. Presence of major vascular invasion on dynamic CT or dynamic MRI

     ① an intraluminal filling defect adjacent to the primary tumor in portal vein, hepatic vein, and/or inferior vena cava

     ② an enhancement of the filling defect on arterial phase and a washout on portal/delayed phases.
  6. Sorafenib naïve or sorafenib experienced
  7. Child-Pugh class A
  8. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1
  9. Life expectancy of at least 16 weeks
  10. Adequate hematologic and hepatic function (should be obtained within 14 days prior to screening:

      * Hemoglobin ≥ 9.0 g/dL

        * Absolute neutrophil count (ANC) ≥ 1,000/mm3 ③ Platelet count ≥ 50,000/μL

          * Total bilirubin < 2.5 mg/dL

            * Serum albumin >2.8 g/dL ⑥ Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 × upper limit of normal (ULN) ⑦ Prothrombin time in INR ≤ 1.8 × ULN ⑧ Serum creatinine ≤ 1.5 mg/dL
  11. Women of childbearing potential and men must agree to use highly efficient contraception since signing of the IC form until at least 5 months (women) and 7 months (men) after the last study drug administration.

Exclusion Criteria:

* Patients with HCC meeting all of following criteria;

  1. Receipt of 2 or more prior systemic therapies for advanced HCC. Additional prior systemic therapies used as adjuvant or local therapy are allowed.
  2. Any type of anticancer agent (including investigational) within 2 weeks before enrollment
  3. Having active brain metastasis or leptomeningeal metastasis
  4. Moderate to severe or intractable ascites
  5. A history or presence of hepatic encephalopathy
  6. Presence of active bacterial infection
  7. Untreated active chronic hepatitis B
  8. History of portal hypertension with bleeding within the past 6 months
  9. Prior liver transplant
  10. Uncontrolled severe medical comorbidity
  11. Other malignant disease (a history of treated malignancy -other than HCC- is allowable if the patient's malignancy has been in complete remission, off chemotherapy and without additional surgical intervention, during the preceding two years)
  12. Current or past history of hypersensitivity to nivolumab

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | through study completion, an average of 2.5 year.
  Progression-free survival (PFS) is defined as the time from the date of treatment initiation to the date of the first observation of progressive disease (PD) by independent radiologic review according to RECIST criteria (version 1.1) or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Joong Won Park, Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Korea, Seoul, South Korea

REFERENCES:
- [Derived] Kim BH, Park HC, Kim TH, Koh YH, Hong JY, Cho Y, Sinn DH, Park B, Park JW. Concurrent nivolumab and external beam radiation therapy for hepatocellular carcinoma with macrovascular invasion: A phase II study. JHEP Rep. 2023 Dec 21;6(4):100991. doi: 10.1016/j.jhepr.2023.100991. eCollection 2024 Apr. PMID 38463541